CLINICAL TRIAL: NCT00380926
Title: Anti-Inflammatory Effect of Polyunsaturated Fatty Acids in Allergic Asthma After Allergen Challenge
Brief Title: Fish Oil and Asthma in House Dust Mite Allergy
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Johann Wolfgang Goethe University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ZAFES-2004-07
Record Dates: First submitted 2006-09-25; First posted 2006-09-27 (Estimated); Last update posted 2006-09-29 (Estimated); Status verified 2006-09

CONDITIONS: Allergic Asthma; Bronchial Inflammation; House Dust Mite Allergy
Keywords: polyunsatturated fatty acids; nutrition; low-dose allergen challenge; exhaled nitric oxide
MeSH Terms: conditions — Dust Mite Allergy | interventions — Fish Oils

INTERVENTIONS:
Drug: polyunsatturated fatty acids (fish oil)

SUMMARY:
Native populations consuming high amounts of fish suffer less from allergic diseases. The purpose of this study is to determine whether polyunsaturated fatty acids (fish oil) might have a disease modifying influence on asthmatics sensitized to house dust mite.

DETAILED DESCRIPTION:
Most asthmatics suffer from mild disease and non pharmacologic intervention would be beneficial for the majority of these subjects. We investigated the anti-inflammatory potential of polyunsaturated fatty acids (PUFA) in allergic asthma.

In our parallel, double-blinded study, 23 patients allergic to house dust mite were randomly assigned to dietary supplementation with a PUFA enriched fat blend or placebo for five weeks. The verum contained eicosapentaenoic acid (EPA) 450 mg/day, docosahexaenoic acid 180 mg/day, stearidonic acid 60mg/day, and gamma-linolenic acid 60 mg/day; the placebo consisted of mainly unsaturated and monosaturated fatty acids. After three weeks, the patients were challenged with low doses of inhalative house dust mite allergen for two weeks.

Following parameters were determined during low-dose allergen exposure in both groups: exhaled NO (eNO) as a marker of bronchial inflammation, clinical symptoms, FEV1, beta-agonist usage, and bronchial hyperreactivity, sputum eosinophils and sulfoleucotrienes. Compliance with the study protocol was controlled by the determination of PUFAs in plasma and erythrocytes.

ELIGIBILITY:
Inclusion Criteria:

* allergic sensitization to house dust mite as proven by skin test and specific IgE
* normal lung function, episodic asthma

Exclusion Criteria:

* history of hypersensitization towards fish oil, chronic illness, pregnancy

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23
Dates: Start 2004-04; Study Completion 2004-11

PRIMARY OUTCOMES:
lung function, symptom score,exhalative nitric oxide, metacholine testing

SECONDARY OUTCOMES:
sulfoleucotriens, eosinophilic cationic protein, sputum eosinophils, safety lab parameters (clinical chemistry, hematology, hemostasis)

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Stefan Zielen, M.D., Principal Investigator — Goethe University, Dpt of Pulmonology/Allergy

REFERENCES:
- [Background] Horrobin DF. Low prevalences of coronary heart disease (CHD), psoriasis, asthma and rheumatoid arthritis in Eskimos: are they caused by high dietary intake of eicosapentaenoic acid (EPA), a genetic variation of essential fatty acid (EFA) metabolism or a combination of both? Med Hypotheses. 1987; 22(4):421-8. Stephensen CB. Fish oil and inflammatory disease: is asthma the next target for n-3 fatty acid supplements? Nutr Rev 2004; 62:486-489 Woods RK, Thien FC, Abramson MJ. Dietary marine fatty acids (fish oil) for asthma in adults and children. Cochrane Database Syst Rev2002; CD001283 Dry J, Vincent D. Effect of a fish oil diet on asthma: results of a 1-year double-blind study. Int Arch Allergy Appl Immunol 1991; 95:156-157 Stenius-Aarniala B, Aro A, Hakulinen A, Ahola I, Seppala E, Vapaatalo H. Evening primrose oil and fish oil are ineffective as supplementary treatment of bronchial asthma. Ann Allergy 1989; 62:534-537 Mickleborough TD, Lindley MR, Ionescu AA, Fly AD. Protective effect of fish oil supplementation on exercise-induced bronchoconstriction in asthma. Chest 2006; 129:39-49